CLINICAL TRIAL: NCT05087537
Title: Effect of Concomitant Bladder Neck Incision and Urethral Valve Ablation on Surgical Re-intervention Rate for Patients With Posterior Urethral Valve : A Randomized Controlled Trial
Brief Title: Effect of Concomitant Bladder Neck Incision and Urethral Valve Ablation on Surgical Re-intervention Rate for Patients With Posterior Urethral Valve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUV , BNI
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Pediatric Disorder; Hydronephrosis in Children; Hydronephrosis, Secondary; Hydronephrosis Congenital; Bladder-Neck; Obstruction, Congenital; Urethral Valve; Renal Function Disorder
Keywords: PUV; BNI; Urethral valve; Valve ablation; Bladder dysfunction
MeSH Terms: conditions — Hydronephrosis; Neoplasm Metastasis; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valve ablation (Active Comparator): Valve ablation
  Interventions: Procedure: Valve ablation
- Valve ablation and bladder neck incision (Active Comparator): Valve ablation and bladder neck incision
  Interventions: Procedure: Valve ablation and bladder neck incision

INTERVENTIONS:
Procedure: Valve ablation — Valve ablation
  Arms: Valve ablation
Procedure: Valve ablation and bladder neck incision — Valve ablation and bladder neck incision
  Arms: Valve ablation and bladder neck incision

SUMMARY:
To determine the short-term effects of concurrent valve ablation and bladder neck incision on re-intervention rate for patients with posterior urethral valve.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are less than 12 years of age with presenting to the Mansoura University Urology and Nephrology Center with the diagnosis of PUV will be s creended for eligibility

Exclusion Criteria:

* Patients with other conditions that can potentially affect lower and upper urinary tract functions
* Patients who were treated with urinary diversion as vesicostomy or cutaneous ureterostomy.
* Patients who had primary treatment of posterior urethral valve ablation at other hospitals.

Max Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — males less than 12 years old
Enrollment: 62 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
compare numbers of reintervention between groups | 1 year
  assessed by calculating the number of patients needed surgical reintervention per total number of patients in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and nephrology center, Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No